CLINICAL TRIAL: NCT03332069
Title: A Phase III Randomised Trial Investigating the Benefits of the Addition of Modulated Electro-hyperthermia to Chemo-radiation for Cervical Cancer in HIV Positive and Negative Women in South Africa
Brief Title: Modulated Electro-Hyperthermia Plus Chemo-radiation for Locally Advanced Cervical Cancer Patients in South Africa
Acronym: mEHT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jeffrey Kotzen (Other)
Collaborators: National Research Foundation of South Africa (Other); NTP Radioisotopes SOC Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Jeffrey Kotzen, Senior Radiation Oncologist, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LACC-OT
Record Dates: First submitted 2017-08-27; First posted 2017-11-06 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Cervical Cancer
Keywords: Hyperthermia; cervix; HIV
MeSH Terms: conditions — Uterine Cervical Neoplasms; Hyperthermia | interventions — Radiotherapy; Cisplatin; Drug Therapy; Brachytherapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Clinicians conducting follow up evaluations, radiographers and nuclear medicine physicians reporting on the PET/CT investigations are unaware of the group that the participants have been assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study (Experimental): 50 Gy external beam radiation administered in fractions of 2 Gy 3 Doses of 8 Gy High Dose Rate brachytherapy up to 3 doses of 80mg/m2 of Cisplatin 10 modulated electro-hyperthermia treatments (55 minutes at a maximum of 150W)
  Interventions: Device: Modulated electro-hyperthermia; Radiation: External beam radiation; Drug: Cisplatin; Radiation: Brachytherapy
- Control (Active Comparator): 50 Gy external beam radiation administered in fractions of 2 Gy 3 Doses of 8 Gy High Dose Rate brachytherapy up to 3 doses of 80mg/m2 of Cisplatin
  Interventions: Radiation: External beam radiation; Drug: Cisplatin; Radiation: Brachytherapy

INTERVENTIONS:
Device: Modulated electro-hyperthermia — Modulated electro-hyperthermia device used is the EHY 2000 by Oncotherm GmbH
  Other Names: Oncothermia; Nanothermia
  Arms: Study
Radiation: External beam radiation
  Other Names: Radiotherapy
Drug: Cisplatin
  Other Names: Chemotherapy
Radiation: Brachytherapy — High Dose Rate
  Other Names: Radiation therapy

SUMMARY:
This is a phase III randomised clinical trial. The aim is to investigate the clinical effects of the addition of modulated electro-hyperthermia (mEHT) to standard treatment protocols (chemoradiotherapy, CRT) for Human Immunodeficiency Virus (HIV) positive and negative locally advanced cervical cancer patients (LACC). SAMPLE: The investigators aim to enrol 236 HIV negative and HIV positive women with LACC, FIGO (Fédération Internationale de Gynécologie et d'Obstétrique) Stages IIB (distil) to stage III. Participants will be randomly assigned to a control group (N=118) and a study group (N=118). METHODOLOGY: Randomisation is based on age, stage and HIV. Participants from both groups will receive the standard treatment for cervical cancer at the hospital at the Charlotte Maxeke Johannesburg Academic Hospital in South Africa: Up to three doses of 80mg/m2 cisplatin, administered three weeks apart; 50Gy external beam radiation (EBR) in fractions of 2Gy; Three doses of 8Gy High Dose Rate (HDR) brachytherapy. The study group will have two 55 minute mEHT treatments per week, at 130W, directly before the EBR using the EHY 2000 Device. OUTCOMES: 1) Determine the local disease control after treatment at 6 months using a Positron Emission Tomography (PET) and computerised tomography (CT) scans. 2) Determine the progression-free survival (PFS) at 6, 12, 18 and 24 months after the last treatment date. PFS will be assessed in all registered participants, regardless of completion (Intent to Treat-ITT) as well as only in the subset of participants who complete the prescribed CRT. 3) Overall survival at two years will be assessed. 4) To evaluate the adverse events associated with mEHT. 5) The effect of mEHT on chemotherapy and radiotherapy tolerability and toxicity will be evaluated. 6) The quality of life of enrolled participants will be assessed before, at 6 weeks, and at 3, 6, 9, 12, 18 and 24 months after completion of therapy using the EORTC (European Organisation for Research and Treatment of Cancer) and EuroQoL forms. 7) To evaluate the economic viability of the addition of mEHT to standard treatment protocols for LACC. 8) The effect, if any, of mEHT treatments on the HIV disease status of HIV positive patients will be assessed by the presence of Autoimmune Deficiency Syndrome (AIDS) defining illnesses before and after treatment. 9) The cancer recurrence patterns will be described and compared in all the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants (who have been adequately clinically staged by standard clinical guidelines) with biopsy proven primary, untreated, histologically confirmed invasive squamous and aden-squamous cell carcinoma of the uterine cervix, FIGO (Fédération Internationale de Gynécologie et d'Obstétrique) stages advanced IIB (invasion of the distal half of the parametrium), IIIA and IIIB.
2. HIV positive participants will be accepted.
3. The following laboratory tests will be done prior to enrolment in the study and the values must be in the following ranges:

   * Haemoglobin >10 g/dL;
   * Platelet count >150/mm3;
   * Absolute neutrophil count (ANC) >3000/mm3
   * Creatinine clearance>60 mL/min
   * Liver function tests
4. Females between the ages of 18 and 70 years.
5. Ability to understand and the willingness to sign a written informed consent document.
6. Eastern Cooperative Oncology Group (ECOG) score of not more than 2.
7. Participants of childbearing potential must have a negative urine or serum pregnancy test prior to enrolment and use an effective form of contraception (e.g. barrier contraception, highly effective hormonal contraception).
8. At the investigators' discretion, participants must be suitable for treatment with radical intent using concurrent chemotherapy and pelvic radiation. Subjects who undergo emergency RT in the form of brachytherapy for haemostasis, prior to enrolment will be allowed to be screened and enrolled provided they meet all other eligibility criteria.
9. Life expectancy of greater than 12 months.
10. Participants must have a body mass index (BMI) that is within normal ranges.

    -

Exclusion Criteria:

1. Participants who have undergone hysterectomy.
2. Exclude para-aortic lymph involvement on planning CT (without contrast)
3. Patients with life-threatening AIDS defining illnesses (other than cervical carcinoma) will be excluded, as will patients with a CD4 count < 200/µL and not on ARVs.
4. Patients with acute active (such as tuberculosis or malaria), serious, uncontrolled infections will be excluded.
5. Participants will be excluded if there is evidence of resistance to antiretroviral therapy (i.e. HIV viral load > 400 copies/mL despite combination antiretroviral therapy for at least 4 months).
6. Prior invasive malignancy other than cervical cancer, diagnosed within the past 24 months, excluding in situ anal dysplasia or carcinoma in situ, non-melanoma skin carcinoma, or Kaposi's sarcoma that has not required systemic chemotherapy within the past 24 months.
7. Pregnant or breast-feeding women.
8. A medical or psychiatric illness that prevents the participant from being able to sign an informed consent or would affect the participant's ability to comply with the protocol stipulations.
9. Participants with circumstances that will not permit completion of the study or required follow-ups. For instance if travel to and from treatment site is an issue.
10. Participants with carcinoma of the cervical stump.
11. Participants with a history of cardiovascular disease manifested as

    1. History of myocardial infarction
    2. Unstable angina
    3. Currently taking medication for treatment of angina
    4. History of coronary artery bypass surgery
12. Participants with contraindications to modulated electro-hyperthermia treatment:

    1. Pace makers and other implanted devices which rely on current and charges.
    2. Large metal implants, such as hip replacements.
    3. Inability to feel temperature in the region.
    4. Inability to express or vocalise discomfort or heat at the treatment site.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2014-01-09 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in Local Disease Control | 6 months post treatment
  Assessed by PET/CT using the RESIST/PERSIST criteria: complete response, complete metabolic response, partial response, stable disease, progressive disease.

SECONDARY OUTCOMES:
Progression Free Survival | 24 months post treatment
  To determine the progression-free survival (PFS) at 6, 12, 18 and 24 months after the last treatment date.
  1. Determine PFS in all registered participants, regardless of completion (Intent To Treat-ITT)
  2. Determine PFS in the subset of participants who complete the prescribed chemo-radiotherapy
2 Year Survival | 24 months post treatment
  Determine the overall survival at two years and the cause of death (i.e. cancer-related, HIV-related, treatment related or other).
Incidence of Adverse Events Attributed to mEHT as assessed by CTCAE version 4.0 | 6 months post treatment
  To evaluate the adverse events that can be directly attributed to mEHT treatments.
Incidence of Treatment Related Adverse Events Attributed to Cisplatin as assessed by CTCAE version 4.0 | Up to 3 months post treatment completion
  The incidence of treatment-emergent adverse events which can be attributed to Cisplatin in each arm will be compared in order to identify any potential effect of mEHT on the frequency and severity of adverse events attributed to Cisplatin.
Number of participants with Early Treatment Related Adverse Events as assessed by CTCAE version 4.0 | Up to 6 months post treatment completion
  The incidence of early toxicity symptoms (graded using the CTCAE version 4 criteria) associated with radiotherapy in each arm of the study will be compared to identify any potential effect of the mEHT on the incidence and severity of early toxicity.
Number of participants with Late Treatment Related Adverse Events as assessed by CTCAE version 4.0 | Up to 24 months post treatment completion
  The incidence of late toxicity symptoms (graded using the CTCAE version 4 criteria) associated with radiotherapy in each arm of the study will be compared to identify any potential effect of the mEHT on the incidence of late toxicity in the sample group.
Visual Analogue Scale On the EuroQoL EQ-5D-5L form | Up to 24 months post treatment completion
  To evaluate the changes from baseline value at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Visual Analogue Scale on the EuroQoL EQ-5D-5L form
Mobility On the EuroQoL EQ-5D-5L form | Up to 24 months post treatment completion
  To evaluate the changes from baseline value at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of Mobility on the EuroQoL EQ-5D-5L form
Self-Care On the EuroQoL EQ-5D-5L form | Up to 24 months post treatment completion
  To evaluate the changes from baseline value at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of Self-Care on the EuroQoL EQ-5D-5L form
Usual Activities On the EuroQoL EQ-5D-5L form | Up to 24 months post treatment completion
  To evaluate the changes from baseline value at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of Usual Activities on the EuroQoL EQ-5D-5L form
Pain/Discomfort On the EuroQoL EQ-5D-5L form | Up to 24 months post treatment completion
  To evaluate the changes from baseline value at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of Pain/Discomfort on the EuroQoL EQ-5D-5L form
Anxiety/Depression On the EuroQoL EQ-5D-5L form | Up to 24 months post treatment completion
  To evaluate the changes from baseline value at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of Anxiety/Depression on the EuroQoL EQ-5D-5L form
Score on the EORTC-QLQ 30 for Global Health Status | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Global Health Status
Score on the EORTC-QLQ 30 for Physical Functioning | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Physical Functioning
Score on the EORTC-QLQ 30 for Role Functioning | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Role Functioning
Score on the EORTC-QLQ 30 for Emotional Functioning | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Emotional Functioning
Score on the EORTC-QLQ 30 for Cognitive Functioning | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Cognitive Functioning
Score on the EORTC-QLQ 30 for Social Functioning | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Social Functioning
Score on the EORTC-QLQ 30 for Fatigue | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Fatigue
Score on the EORTC-QLQ 30 for Nausea and Vomiting | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Nausea and Vomiting
Score on the EORTC-QLQ 30 for Pain | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Pain
Score on the EORTC-QLQ 30 for Dyspnoea | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Dyspnoea
Score on the EORTC-QLQ 30 for Insomnia | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Insomnia
Score on the EORTC-QLQ 30 for Appetite Loss | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Appetite Loss
Score on the EORTC-QLQ 30 for Constipation | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Constipation
Score on the EORTC-QLQ 30 for Diarrhoea | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Diarrhoea
Score on the EORTC-QLQ 30 for Financial Difficulties | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Financial Difficulties
Score on the EORTC-QLQ 24 for Symptom Experiences | Up to 24 months post treatment completion
  To evaluate the changes from baseline scores at set time points (6 weeks, 3 months, 6 months, 9 months, 12 months,18 months, 24 months) of the Score on the EORTC-QLQ 30 for Symptom Experiences

CONTACTS AND LOCATIONS:
Overall Officials: Carrie A Minnaar, Msc, Study Chair — Student - PhD Candidate; Jeffrey A Kotzen, MBBCH, Principal Investigator — Senior Radiation Oncologist; Ans Baeyes, PhD, Study Chair — Head of Department of Radiobiology
Locations (1):
- Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fiorentini G, Szasz A. Hyperthermia today: electric energy, a new opportunity in cancer treatment. J Cancer Res Ther. 2006 Apr-Jun;2(2):41-6. doi: 10.4103/0973-1482.25848. PMID 17998673
- [Background] van der Zee J, Gonzalez GD. The Dutch Deep Hyperthermia Trial: results in cervical cancer. Int J Hyperthermia. 2002 Jan-Feb;18(1):1-12. doi: 10.1080/02656730110091919. PMID 11820462
- [Derived] Minnaar CA, Kotzen JA, Naidoo T, Tunmer M, Sharma V, Vangu MD, Baeyens A. Analysis of the effects of mEHT on the treatment-related toxicity and quality of life of HIV-positive cervical cancer patients. Int J Hyperthermia. 2020;37(1):263-272. doi: 10.1080/02656736.2020.1737253. PMID 32180481
- [Derived] Minnaar CA, Kotzen JA, Ayeni OA, Naidoo T, Tunmer M, Sharma V, Vangu MD, Baeyens A. The effect of modulated electro-hyperthermia on local disease control in HIV-positive and -negative cervical cancer women in South Africa: Early results from a phase III randomised controlled trial. PLoS One. 2019 Jun 19;14(6):e0217894. doi: 10.1371/journal.pone.0217894. eCollection 2019. PMID 31216321